CLINICAL TRIAL: NCT02920203
Title: Genetic Autopsy and Sudden Death of Young Subject
Brief Title: Genetic Autopsy and Sudden Death
Acronym: AGEMOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pathology department and forensic Institute, Raymond Poincaré hospital, Garches (Unknown); Referal Center for Inherited cardiac diseases, Pitié Salpêtrière Hospital, Paris (Unknown); Pitié-Salpêtrière Hospital (Other); Clinical research Unit, Ambroise Paré Hospital, Boulogne Billancourt (Unknown); Cardiogenetic and molecular and cellular myogenetic functionnal unit Pitié Salpêtrière hospital, Paris (Unknown); Molecular and medical Virology Laboratory, Medical School, Reims (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI 13007
Record Dates: First submitted 2016-09-07; First posted 2016-09-30 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Sudden Death
Keywords: Sudden unexpected death; young subjects; molecular genetic autopsy; sequencing
MeSH Terms: conditions — Death, Sudden

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Heart and spleen tissue (from autopsy)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- index cases group: unexpected sudden death cases recruited by forensic institutes or pathology departements
  Interventions: Genetic: Heart and spleen tissue
- first degree relatives group: Relatives enrolled of unexpected sudden death index cases

INTERVENTIONS:
Genetic: Heart and spleen tissue — genetic sequencing
  Groups: index cases group

SUMMARY:
The purpose of the study is to better identify hereditary cardiac causes of sudden unexpected death in young subjects through Next-Generation Sequencing of autopsy tissue

DETAILED DESCRIPTION:
Monitoring :

For index cases group, all the data will be monitored. For the relatives group, only the informed consent will be monitored

Statistical analysis :

* Evaluate the additional elucidation rate of unexpected sudden death
* Evaluate causes obtained by Next Generation Sequencing (NGS) ( in comparison with conventional autopsy (macroscopic and / or microscopic)
* Descriptive study of the causes of sudden unexpected death, identified hereditary cardiac causes percentages compared via various diagnostic approaches
* Cost-effectiveness analysis

Data Management :

A database is created for the AGEMOS study with control of the discrepancies. All the index cases' data entered in the data base will be double checked

ELIGIBILITY:
Index cases :

Inclusion Criteria:

* Subjects of more than 2 years old and less than 41 years old
* Sudden unexpected death from natural and nontraumatic causes
* Macroscopic autopsy performed within 72 hours after death and without signs of body decomposition
* No extracardiac obvious causes, including toxicological analysis when available
* No significant coronary cause after autopsy (such as tight coronary stenosis, congenital abnormality of the arteries, coronary vasculitis)
* Informed consent of the close relation (family/reliable person) and / or legal representative

Relatives :

Inclusion Criteria:

* To be a first degree relative (parents, sister, brother, child) of a deceased subject included in the AGEMOS study and accept to perform medical examination and transmit results of examination

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Index cases enrolled: series of consecutive and exhaustive cases recruited by forensic institutes or pathology departements Relatives enrolled: as many as possible during the recruitment period
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of sudden death elucidation rate obtained by high throughput sequencing (NGS) versus conventional autopsy (macroscopic and / or microscopic) | 27 months
  Aim is to determine if elucidation rate of unexpected sudden death causes obtained by high throughput sequencing (NGS) is significantly better than conventional autopsy (macroscopic and / or microscopic) alone.
  Inclusion of a series of 100 consecutive and exhaustive cases (index cases) recruited by forensic institutes or pathology departements.
  Determine the rate of sudden death elucidation after NGS (after targeted capturing of 100 genes responsible for inherited cardiac diseases, including cardiomyopathy and electrical diseases) and comparison of sudden death elucidation rate obtained with conventional autopsy (macroscopic and microscopic) by chi 2 analysis.

SECONDARY OUTCOMES:
Describe the epidemiology of causes of sudden death | 27 months
  Inclusion of a serie of consecutive and exhaustive subjects recruited by forensic institutes or pathology departements.
  Determination all the causes of death after conventional autopsy (unnatural, toxicological, non-cardiovascular, vascular, cardiological and coronary, cardiological and non-coronary causes such as cardiomyopathies & myocarditis, no cause identified Descriptive analysis. All quantitative data will be analyzed with the average, standard deviation and median.
  Frequencies and Clopper-Pearson confidence interval of 95% will be provided
Comparison of elucidation rates of cause of sudden death including systematic cardiac screening in relatives | 39 months
  Aim is to determine the impact of systematic family cardiac screening in the understanding of sudden deaths Comparison of elucidation rates of cause of sudden death according to three methods:
  i) identification of a hereditary heart disease via the systematic cardiac screening performed in relative; ii) by the conventional autopsy; iii) by sequencing NGS analysis; Statistics: test of McNemar (mated series). The threshold for level of statistical significance is chosen at 5 %.
Medico-economic modeling of the various diagnostic approaches | 39 months
  Cost-effectiveness modeling evaluation of medical and economic impact of the genetic molecular autopsy, efficacy being estimated by years of life saved in the family

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy Lorin de la Grandmaison, Pr, Principal Investigator — Assistance Publique Hoptiaux de Paris; Philippe Charron, MD, PhD, Study Director — +33 (0)1 42 16 13 47
Locations (1):
- Raymond Poincaré hospital, Garches, France

IPD SHARING:
Plan to Share IPD: No